CLINICAL TRIAL: NCT06732297
Title: Stronger Family Through Art Therapy: a Mixed Methods Programme Evaluation Study
Acronym: SFAT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanyang Technological University (Other)
Collaborators: The Red Pencil Singapore (Unknown); National Council Of Social Service, Singapore (Other); The Majurity Trust (Unknown)
Responsible Party: Principal Investigator, Andy Hau Yan Ho, PhD, EdD, Professor, Nanyang Technological University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: IRB-2024-821
Record Dates: First submitted 2024-12-10; First posted 2024-12-13 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Vulnerable Families
Keywords: Vulnerable families; art therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Immediate Treatment Group (Experimental): Participants in the immediate treatment group will undergo the intervention after baseline assessment and randomization. The intervention consists of 1.5-hour art-therapy sessions which happen every week for 10 weeks. The topics of intervention sessions include building rapport, emotional expression & regulation, self-care, communication & collaboration, and reflection & community.
  Interventions: Behavioral: dyadic art therapy intervention for parent-child relationship in vulnerable families
- Waitlist Control Group (Other): Participants in the waitlist control group will undergo the intervention after participants in the immediate treatment group complete the intervention. Participants in the two group undergo the same intervention.
  Interventions: Behavioral: dyadic art therapy intervention for parent-child relationship in vulnerable families

INTERVENTIONS:
Behavioral: dyadic art therapy intervention for parent-child relationship in vulnerable families — The Stronger Family Through Art Therapy (SFAT) is a dyadic art therapy intervention developed to improve the parent-child relationship in vulnerable families. Service users of the SFAT programme will receive a progressive support from workshops, dyad art therapy, and an innovative art-based self-care tool developed with a multidisciplinary team to meet the needs of enhancing family communication and strengthening emotional bonding.

SUMMARY:
The current research aims to evaluate the effectiveness and feasibility of the Strong Family Through Art Therapy (SFAT) programme, which was developed to improve the parent-child relationship in vulnerable families. The main questions it aims to answer are:

1. Is the programme effective in enhancing quality of life and family resilience among parents?
2. Is the programme effective in enhancing quality of life among children?
3. Is the programme feasible and acceptable for large scale implementation in Singapore?

Researchers will compare participants before and after they take the programme and compare participants who take the programme with participants with participants who have not yet taken the programme to see if the programme is effective in benefiting participants. Researchers will also invite participants to discuss together and interview art therapists to see if the programme is feasible and acceptable.

Participants will

1. Take the 10-week SFAT programme
2. Complete assessment survey for 3 times
3. Attend a focus group discussion

DETAILED DESCRIPTION:
The current research aims to evaluate the effectiveness and feasibility of the Strong Family Through Art Therapy (SFAT) programme, which was developed to improve the parent-child relationship in vulnerable families. Service users of the SFAT programme will receive a progressive support from workshops, dyad art therapy, and an innovative art-based self-care tool developed with a multidisciplinary team to meet the needs of enhancing family communication and strengthening emotional bonding. The current research utilizes a pragmatic mixed method research paradigm to evaluate the programme. For the quantitative component, a single-site, open label, Waitlist Randomized Control Trial (RCT) design, comprising two arms: (i) treatment group and (ii) waitlist control group, will be adopted to evaluate the efficacy of the Strong Family Through Art Therapy (SFAT) for improving quality of life and family resilience among parents and children. For the qualitative component, an embedded qualitative focus group evaluation study with participants who complete the SFAT programme, together with analysis of intervention session evaluation forms completed by the RPS art therapists who conduct the SFAT programme, will be conducted to evaluate programme acceptability and feasibility. After signing the informed consent form, the recruited family(consisting of one parent and one to three children dyads) will be asked to complete a baseline assessment before randomization and the start of the SFAT programme [T1]. Treatment group participants will then undergo an 10-week SFAT programme conducted by the RPS clinical team, complete an immediate post-intervention assessment [T2], with a final follow-up assessment at 20-weeks [T3]. The waitlist control group will complete a pre-intervention assessment before start of the SFAT programme at 10-weeks [T2], then undergo the same 10-week SFAT programme conducted by the RPS clinical team and complete an immediate post-intervention assessment at 20-weeks [T3]. Moreover, selected participants will be invited to take part in an acceptability focus group study after T3 assessments. Post-session evaluation forms will also be completed by RPS art therapists after session completion. Figure 1 details the study procedures.

ELIGIBILITY:
Inclusion Criteria:

* the caregiver (including parents, grandparents, family members or foster parents who perform the main caretaking responsibilities of the children taking part in SFAT) of a young child who can communicate in English and provide informed consent
* the child is aged 7-14 years and can communicate in English
* the family have one or more of the following identified challenges: (1) caregiver stress such as finances, household management, work and childcare arrangements, (2) caregiver struggles to find time for self-care and quality time with children, (3) caregiver has minimal understanding of the psychological and emotional needs of their children, (4) children face difficulties with emotional regulation and anger management
* caregivers and children are from low-income families who receive financial assistance under the CHAS Blue card, ComCare financial assistance, and/or the MOE Financial Assistance Scheme

Exclusion Criteria:

* individuals who are suffering from depression or other major mental health conditions that would render their participation highly disruptive to others in a group setting, and/or cannot provide informed consent. Families will also be excluded if they are currently unstable (i.e. circumstances related to abuse/neglect), and/or have high risk of suicidal and self-harm behaviours. In the cases that individuals referred to the programme are not eligible, the partner organisations will assess their needs and refer them to programmes based on these needs.
* participant is unable to provide informed consent

Ages: 7 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Self-rated quality of life for caregivers | From enrollment to the end of assessment at 20 weeks
  The primary outcome will be assessed by the World Health Organization Quality of life Brief Scale (WHOQOL-BREF) [WHO, 1997]. The WHOQOL-BREF comprises 26-items rated on a 5-point Likert scale and clustered into the four subscales of physical health, psychological health, social relationships, and environmental health. The WHOQOL-BREF possesses strong internal validity, reliability, and cross-cultural applicability.
Self-rated quality of life for children | From enrollment to the end of assessment at 20 weeks
  The primary outcome will be assessed by the KIDSCREEN-30 tool [Ravens-Sieberer, U., et al., 2013]. The KIDSCREEN-30 comprises of 30 items rated on a 4-point visual Likert scale and clustered into the 8 domains of physical wellbeing, psychological wellbeing, moods and emotions, autonomy and parent relation, financial resources, social support and peers, school environment and social acceptance. KIDSCREEN30 possesses strong internal validity, reliability, and cross-cultural applicability.

SECONDARY OUTCOMES:
Self-rated family resilience for caregivers | From enrollment to the end of assessment at 20 weeks
  The secondary outcome will be assessed by the Walsh Family Resilience Questionnaire (WFRQ) [Walsh, 2016]. The WFRQ comprises 32 items rated on a 5- point Likert Scale and clustered into the 3 subscales of belief systems, organisational pattens, and communication/problem solving. The WFRQ possesses strong internal validity, reliability, and cross-cultural applicability

CONTACTS AND LOCATIONS:
Locations (1):
- The Red Pencil Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No